CLINICAL TRIAL: NCT05756764
Title: Pilot Study of the Effect of Weight Loss by Pharmacotherapy on Chronic Pro-tumor Inflammatory Cells
Brief Title: Anti-obesity Pharmacotherapy and Inflammation
Status: Active, not recruiting | Type: Observational
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: Tulane University (Other); Pennington Biomedical Research Center (Other); Ochsner Health System (Other)
Responsible Party: Principal Investigator, Maria Sanchez-Pino, Ph.D., Assistant Professor, Louisiana State University Health Sciences Center in New Orleans
Other Study IDs: U24DK132740-5053; U24DK132740 (NIH)
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Obesity
Keywords: Inflammation; Dyslipidemia; Metabolic syndrome
MeSH Terms: conditions — Obesity; Inflammation; Dyslipidemias; Metabolic Syndrome | interventions — semaglutide; Glucagon-Like Peptide-1 Receptor; Qsymia; Phentermine; Tirzepatide; Topiramate; Diethylpropion; Naltrexone; Bupropion; bupropion hydrochloride, naltrexone hydrochoride drug combination; Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood will be obtained from participant subjects. Collection of serum, plasma, and isolation of leukocytes will be used for study aims and storage (-80 degrees).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with obesity on pharmacotherapy: Before initiation of pharmacotherapy (as part of the standard-of-care treatment) and 6 months after initiated medication
  Interventions: Drug: Semaglutide; Drug: Phentermine-Topiramate combination; Drug: Phentermine; Drug: Tirzepatide; Drug: Topiramate; Drug: Diethylpropion; Drug: Naltrexone/Bupropion; Drug: Liraglutide

INTERVENTIONS:
Drug: Semaglutide — Medication for weight loss
  Other Names: Glucagon-like peptide-1 receptor (GLP1-R) agonist; Wegovy
Drug: Phentermine-Topiramate combination — Medication for weight loss
  Other Names: Qsymia
Drug: Phentermine — Medication for weight loss
  Other Names: Lomaira; Adipex-P
Drug: Tirzepatide — Medication for weight loss
  Other Names: Mounjaro; Zepbound; GIP/GLP-1 RA
Drug: Topiramate — Medication for weight loss
  Other Names: Topamax; Trokendi XR; Qudexy XR
Drug: Diethylpropion — Medication for weight loss
  Other Names: Tenuate; Diethylcathinone
Drug: Naltrexone/Bupropion — Medication for weight loss
  Other Names: Contrave
Drug: Liraglutide — Medication for weight loss
  Other Names: Saxenda; Victoza; Glucagon-like peptide-1 receptor (GLP1-R) agonist

SUMMARY:
This study evaluates the relationship between weight loss, circulating inflammatory markers and lipids from 24 patients before and after 6 months of pharmacotherapy as a standard of care for anti-obesity treatment

DETAILED DESCRIPTION:
This study aims to determine if weight loss by pharmacotherapy with liraglutide, semaglutide, or phentermine-topiramate promotes the reduction of pro-tumoral inflammatory cells Myeloid-derived suppressor cells (MDSC), simultaneously to the improvement of lipid profile (LDL-Cholesterol, HDL-Cholesterol, triglycerides, and free fatty acids) and concentration in the blood.

Liraglutide, semaglutide, and phentermine-topiramate are FDA-approved medications to treat obesity and obesity-associated comorbidities.

Twenty-four patients undergoing standard of care for anti-obesity treatment at VA Medical Center, and Tulane Center for Clinical Research (TCCR) will be recruited before initiation of pharmacotherapy as part of their standard of care and followed up to 6 months to compare the primary study variables.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI): over 30 kg/m2
* Age: 35 to 60 years old

Exclusion Criteria:

* Taking medications with anti-inflammatory properties like glucocorticoids, prednisone, or non-steroidal anti-inflammatory medications, such as aspirin or Motrin Subjects on medications for long-term weight management such as phentermine-topiramate (Qsymia), orlistat (Xenical), naltrexone-bupropion (Contrave), and the glucagon-like peptide-1 receptor agonists such as liraglutide (Saxenda), and semaglutide (Wegovy).
* Prior history of cancer
* Having any clinical symptoms of systemic inflammation, acute infections such as Coronavirus disease 2019, or chronic diseases such as cancer, tuberculosis, autoimmune disease, and AIDS
* An adult unable to consent
* Prisoner
* Pregnancy or breastfeeding women

Ages: 35 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients with obesity, defined as having a body mass index (BMI) > 30, from New Orleans and its surroundings, scheduled for initiating the anti-obesity treatment with drugs for weight loss as part of their standard-of-care for anti-obesity treatment at Clinics from New Orleans and its surroundings; therefore, the research trial team will not provide the medications. Expect to recruit 50% African American (6 women, 6 men), and 50% White American (6 women, 6 men), as a representative majority of the New Orleans population.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
weight loss | baseline and 24 weeks
  Weight Loss Percentage (Pounds lost divided by starting weight (in pounds) multiplied by 100)
MDSC in peripheral blood | baseline and 24 weeks
  Changes in number of MDSC in blood
Levels of lipids in circulation | baseline and 24 weeks
  Changes in concentration (mg/dL) of each type of lipids: LDL-Cholesterol, triglycerides, and free fatty acids

SECONDARY OUTCOMES:
Systemic inflammation measured by C-reactive protein levels | baseline and 24 weeks
  Changes in concentration (mg/L) of C-reactive protein in serum
Systemic inflammation measured by adipokines levels in circulation | baseline and 24 weeks
  Changes in concentration (pg/mL) of interleukin 6 (IL-6), tumor-necrosis factor alpha (TNFa) and leptin in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Maria D Sanchez-Pino, Ph.D., Principal Investigator — LSU-Health Sciences Center
Locations (2):
- United States (2):
  - LSU Clinical & Translational Research Center (CTRC - - LSUHSC-NO, New Orleans, Louisiana
  - Ochsner Health System - Biospecimen, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: Yes
The investigators will adhere to the NIH Grants Policy on Sharing of Unique Research Resources, including the Sharing of Biomedical Research Resources: Guidelines for Recipients of NIH Grants and Contracts on Obtaining and Disseminating Biomedical Research Resources (NOT-OD-21-013).
  Data dictionaries, statistical analysis code, and de-identified data may be deposited for sharing. Data may include demographic, clinical, anthropometric, outcome measures, and other relevant variables, as allowed by the data-owning organization, consistent with applicable laws and regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data may be deposited into the repository no later than within one year of completing the study period for the award or upon acceptance of the data for publication or public disclosure of study results.
Access Criteria: Deidentified data and supporting information may be shared with investigators and research staff working under a Federal Wide Assurance (FWA) institution and could be used for secondary study purposes after approval of the local Institutional Review Board (IRB)